CLINICAL TRIAL: NCT00920660
Title: A Randomised, Double-blind, Placebo-controlled, Multi-way Crossover Study to Assess the Effects of Single Oral Doses of SRT2104 and Prednisolone on Biomarkers in Blood in Healthy Volunteers
Brief Title: Clinical Study to Assess the Effects of SRT2104 and Prednisolone on Biomarkers in Blood in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 113161
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — SRT2104; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Group (Experimental): Subjects will be required to attend the research unit in a fasted state (at least 10 hours without food) on six separate occasions (treatment visits) during the study. At approximately the same time every morning, subjects will consume a standard, non-high-fat meal (approximately 650 kcal with 30% of calories derived from fat). Test material (per treatment) will be administered within 15-30 minutes following the meal. There will be at least a 7-day washout period between treatment visits.
  During the first five treatment visits, subjects will receive one of the following treatments in the form of 8 capsules: 0.25g SRT2104, 0.5g SRT2104, 1g SRT2104, 2g SRT2104, or placebo.
  During the last treatment visit, subjects will receive 30 mg of open-label prednisolone tablets.
  Interventions: Drug: Placebo; Drug: 0.25g SRT2104; Drug: Prednisolone; Drug: 0.5g SRT2104; Drug: 1g SRT2104; Drug: 2g SRT2104

INTERVENTIONS:
Drug: Placebo — Matching placebo is supplied containing microcrystalline cellulose (Avicel PH 105). Placebo will be administered as eight matched capsules.
Drug: 0.25g SRT2104 — SRT2104 will be supplied as hard gelatin capsules, with each containing 250 mg. The 0.25g SRT2104 treatment visit will be administered as one SRT2104 capsule with 7 placebo capsules. Dosing will take place during one of the 6 treatment visits.
Drug: Prednisolone — During the last treatment period, subjects will receive 30 mg open-label prednisolone.
Drug: 0.5g SRT2104 — SRT2104 will be supplied as hard gelatin capsules, with each containing 250 mg. The 0.5g SRT2104 treatment visit will be administered as two SRT2104 capsules with 6 placebo capsules. Dosing will take place during one of the 6 treatment visits.
Drug: 1g SRT2104 — SRT2104 will be supplied as hard gelatin capsules, with each containing 250 mg. The 1g SRT2104 treatment visit will be administered as four SRT2104 capsules with four placebo capsules. Dosing will take place during one of the 6 treatment visits.
Drug: 2g SRT2104 — SRT2104 will be supplied as hard gelatin capsules, with each containing 250 mg. The 2g SRT2104 treatment visit will be administered as eight SRT2104 capsules. Dosing will take place during one of the 6 treatment visits.

SUMMARY:
The primary purpose of this study is to assess the pharmacodynamic effect of single, oral doses of SRT2104 (250 mg, 500 mg, 1000 mg, 2000 mg) and prednisolone as measured by levels of ex vivo LPS-induced TNF-alpha production in whole blood of healthy adult subjects.

The secondary purposes of this study are to assess the pharmacodynamic effects of single, oral doses of SRT2104 (250 mg, 500 mg, 1000 mg, 2000 mg) and prednisolone (30mg) as measured by levels of IL-6, IL-8 and IL-1beta in whole blood of healthy adult subjects. In addition, plasma pharmacokinetics, safety and tolerability of SRT2104 following the administration of single, oral doses of SRT2104 (250 mg, 500 mg, 1000 mg, 2000 mg) in healthy adult subjects will also be assessed. As exploratory endpoints, transcriptomic profiles, biomarker exploration, and relationships between plasma SRT2104 levels and ex vivo LPS-induced TNF-alpha production may also be examined.

DETAILED DESCRIPTION:
This is a prospective, single center, non-therapeutic clinical study of SRT2104 administered orally as 250 mg capsules. Randomized, double-blind study to evaluate and compare the sensitivity of systemic biomarkers, such as ex-vivo LPS-induced TNF-alpha, IL-6, IL-8, and IL-1beta, to treatment with four-single oral doses of SRT2104 (250 mg, 500 mg, 1000 mg, and 2000 mg), prednisolone (30 mg), and placebo in healthy adult volunteers. Twenty (20) subjects (males and females of non-childbearing potential) aged 18-60, who fulfill the inclusion/exclusion criteria, will be enrolled in this study to achieve a minimum of 15 evaluable subjects. Each subject will participate in 6 treatment periods. For each treatment period subjects will fast for at least 10 hours overnight. After pre-dosing procedures, subjects will consume a standard, non-high-fat (approximately 650 kcal with approximately 30% of calories derived from fat) meal 15-30 minutes prior to receiving test material. During the first five treatment periods, subjects will receive a single dose of SRT2104 or matched placebo; during the last treatment period, subjects will receive 30 mg open-label prednisolone. Assessments will be performed until 24 hours post dose in each treatment period.

Subjects will be asked to sign the informed consent form(s) at the screening visit. If eligible and willing to participate, subjects will enter into the study. Subjects will be required to attend the research unit in a fasted state (at least 10 hours without food) on six separate occasions (treatment visits) during the study. There will be at least a 7-day washout period between treatment visits.

During the first five treatment visits, subjects will receive one of the following five treatments:

A. 250 mg SRT2104 administered as eight oral capsules (one active SRT2104 250 mg capsule + seven placebo capsules) B. 500 mg SRT2104 administered as eight oral capsules (two active SRT2104 250 mg capsules + six placebo capsules) C. 1000 mg SRT2104 administered as eight oral capsules (four active SRT2104 250 mg capsules + four placebo capsules) D. 2000 mg SRT2104 administered as eight oral capsules (eight active SRT2104 250 mg capsules + zero placebo capsules) E. Eight placebo capsules

During the last treatment visit, subjects will receive 30 mg of open-label prednisolone tablets.

Subjects will be required to return to the research unit 24 hours after dosing in each treatment period in order to gather the required PK and PD samples. Subjects will be asked to return to the study center for an End of Study safety assessment 7 to 10 days after the last treatment visit.

ELIGIBILITY:
Inclusion Criteria:

* The study is open to healthy male and female volunteers, 18 to 60 years of age, with hematology, clinical chemistry, electrolytes, serology, and urinalysis tests within normal, allowable limits using normal laboratory values (if out-of-range values result, they must be considered clinically significant by the Investigator to be exclusionary) and performed within 21 days to 1 day of receiving the first dose of test material.
* All male subjects and their female partners must be willing and able to use an acceptable form of double-barrier birth control (hormonal or double barrier method of birth control [condom and occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam, gel, film, cream, or suppository]; true abstinence) for at least 12 weeks after the last treatment dose.
* All female subjects must be of non-childbearing potential. For the purposes of this study, non-childbearing potential is defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory]. [Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use adequate contraception (hormonal or double barrier method of birth control [condom and occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam, gel, film, cream, or suppository]; true abstinence) for the duration of the study dosing and for at least 12 weeks after the last treatment dose, if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method].

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-04-06 (Actual); Primary Completion 2009-06-12 (Actual); Study Completion 2009-06-12 (Actual)

PRIMARY OUTCOMES:
To assess the pharmacodynamic effect of single, oral doses of SRT2104 (250 mg, 500 mg, 1000 mg, and 2000 mg) and prednisolone (30 mg) as measured by levels of ex vivo LPS-induced TNF-alpha production in whole blood of healthy adult subjects. | Duration of treatment periods.

SECONDARY OUTCOMES:
To assess the pharmacodynamic effect of single, oral doses of SRT2104 (250 mg, 500 mg, 1000 mg, and 2000 mg) and prednisolone (30 mg) as measured by levels of IL-6, IL-8 and IL-1beta in whole blood of healthy adult subjects. | Duration of treatment periods.
To assess the plasma pharmacokinetics of SRT2104 following the administration of single, oral doses of SRT2104 (250 mg, 500 mg, 1000 mg, and 2000 mg) in healthy adult subjects. | Duration of treatment periods.
To assess the safety and tolerability of single oral doses of SRT2104 (250 mg, 500 mg, 1000 mg, and 2000 mg) in healthy adult subjects. | Duration of treatment periods.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Merthyr Tydfill, Glamorgan, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 113161 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113161?search=study&study_ids=113161#rs
- Available data/document: Dataset Specification: 113161 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113161 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113161 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113161 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113161 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113161 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113161 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register